CLINICAL TRIAL: NCT00236457
Title: Randomized, Multi-center, Open Label Trial Comparing Risperidone Depot (Microspheres) and Olanzapine Tablets in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study Comparing the Efficacy of Long-acting Injectable Risperidone and Olanzapine Tablets in the Treatment of Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002026
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Schizophrenia; Intramuscular injection; Antipsychotic agents; Long-acting risperidone; Olanzapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to document both short-term, as well as long-term efficacy and safety of a long-acting injectable formulation of risperidone, in comparison with olanzapine for the treatment of patients with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Many schizophrenia patients currently take oral antipsychotic medications daily, but long-acting injectable formulations may eliminate this need for the daily medication. This is an open-label study of a flexible does of a long-acting formulation of risperidone injected into the muscle at 2 week intervals over 12 months in patients with schizophrenia or schizoaffective disorder. A comparator group will receive daily tablets of olanzapine, a psychotropic agent available for the treatment of schizophrenia and schizoaffective disorders. This is a two-part trial. Patients will be titrated to the most effective dose of trial medication during the first 13 weeks and analyzed for short-term efficacy and safety of treatment at Week 13. Patients will be then assessed for maintenance of efficacy, safety, and resource use at Week 52 (second part of study). Efficacy assessments include the Structured Clinical Interview - Positive and Negative Syndrome Scale (SCI-PANSS), overall severity of illness measured by the Clinical Global Impression (CGI) scale, and quality of life assessed by Wisconsin Quality of Life Index (W-QOLI). Safety evaluations include incidence of adverse events, Simpson and Angus Rating Scale for extrapyramidal symptoms, physical examinations, clinical laboratory tests (biochemistry, haematology, and urinalysis), and electrocardiograms (ECGs). The primary study hypothesis is that treatment with long-acting risperidone injected intramuscularly every 2 weeks is not inferior to treatment with daily olanzapine in terms of short-term efficacy and is well tolerated by patients with schizophrenia or schizoaffective disorder. Risperidone injections (25mg or 50mg) every 2 weeks for 12 months. Investigator may decrease or increase dosages (max 50mg) or supplement risperidone injections with risperidone tablets (4mg/day max.). Control group receives olanzapine tablets (5mg) daily, adjusted as necessary (max 20mg).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder according to criteria of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DMS IV)
* Positive and Negative Syndrome Scale (PANSS) total score =>50, indicating at least a minimum level of mental and behavioral disorders
* Recent hospitalization or an episode of psychosis requiring medical intervention
* Body Mass Index (BMI) <=40 (BMI >=30 indicates obesity)

Exclusion Criteria:

* Diagnosis of DMS IV Axis I condition other than schizophrenia or schizoaffective disorder
* History of neuroleptic malignant syndrome, a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness
* Past treatment with clozapine
* Pregnant or nursing females, or those lacking adequate contraception
* Known sensitivity or unresponsiveness to risperidone or olanzapine
* Treatment with a long-acting injectable antipsychotic drug near the time of the trial start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2000-11; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 13 for total score using the Structured Clinical Interview- Positive and Negative Syndrome Scale (SCI-PANSS)

SECONDARY OUTCOMES:
Change from baseline through each visit and at study end (Week 53) for SCI-PANSS total score, SCI-PANSS subscales, Clinical Global Impression (CGI) and Wisconsin Quality of Life Index (W-QOLI). Safety evaluations throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study comparing the efficacy of long-acting injectable risperidone and olanzapine tablets in the treatment of patients with schizophrenia or schizoaffective disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=450&filename=CR002026_CSR.pdf